CLINICAL TRIAL: NCT02509260
Title: A Randomized Controlled Trial of Prevena™ Incisional Negative Pressure Wound Therapy to Reduce Surgical Site Infection in Re-operative Colorectal Surgery
Brief Title: Prevena™ Incisional Negative Pressure Wound Therapy in Re-operative Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, David Liska, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-709
Record Dates: First submitted 2015-07-24; First posted 2015-07-27 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Surgical Site Infection
Keywords: colorectal surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena™ incisional NPWT (Experimental): Prevena wound management system: Post op application of the Prevena™ wound management system will be applied.
  Interventions: Device: Prevena wound management system
- Standard Wound Dressings (Active Comparator): Standard Wound Dressings: Control patients with standard wound dressings will have gauze and tape dressings applied.
  Interventions: Other: Standard wound dressings

INTERVENTIONS:
Device: Prevena wound management system — Patients will have the Prevena wound management system applied post-operatively.
  Arms: Prevena™ incisional NPWT
Other: Standard wound dressings — Control patients with standard wound dressings will have gauze and tape dressings applied
  Arms: Standard Wound Dressings

SUMMARY:
Many strategies have been attempted to reduce SSI rates. The Centers for Medicare and Medicaid Services introduced the Surgical Care Improvement Project infection project with the aim of reducing SSI incidence and morbidity. These measures include prophylactic intravenous antibiotics administered within 1 hour of skin incision, appropriate prophylactic antibiotic selection, discontinuation of prophylactic antibiotics within 24 hours after surgery, appropriate hair removal, and maintenance of perioperative normothermia. Despite the enforcement of these measures through quality reporting and pay-for-performance measures, significant controversy exists as to their overall effectiveness, especially in the high-risk colorectal surgical population. Laparoscopic surgery has been shown to improve SSI rates in the colorectal population; however, not all patients are appropriate candidates for this approach and the inability of promising interventions such as wound edge protection and gentamicin sponges to improve SSI rates following colorectal surgery mandate the investigation of novel techniques.

The aim of the current study is to assess the clinical effectiveness of incisional NPWT to reduce SSI rates in open, re-operative colorectal surgery. The primary endpoint of this study is the occurrence of superficial SSI within 30 days after surgery and the secondary endpoints include length of hospital stay and cost effectiveness.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are a common problem and a significant cause of morbidity in surgical patients. They present a substantial burden to the health care system in the United States and contribute more than 1.6 billion dollars in excess cost and 1 million in extra hospital days in affected patients. SSIs are associated with a multitude of complications including an increased risk of incisional hernia and prolonged hospital stay. Despite optimum surgical care there remains an inability to significantly reduce SSI rates following colorectal surgery and this field represents a critical priority for study. When one examines the control arms of recent high quality randomized controlled trials, the SSI rate following colorectal surgery ranges from 22.0-26.1%, emphasizing the prevalence of this complication.

Many strategies have been attempted to reduce SSI rates. The Centers for Medicare and Medicaid Services introduced the Surgical Care Improvement Project infection project with the aim of reducing SSI incidence and morbidity. These measures include prophylactic intravenous antibiotics administered within 1 hour of skin incision, appropriate prophylactic antibiotic selection, discontinuation of prophylactic antibiotics within 24 hours after surgery, appropriate hair removal, and maintenance of perioperative normothermia. Despite the enforcement of these measures through quality reporting and pay-for-performance measures, significant controversy exists as to their overall effectiveness, especially in the high-risk colorectal surgical population. Laparoscopic surgery has been shown to improve SSI rates in the colorectal population; however, not all patients are appropriate candidates for this approach and the inability of promising interventions such as wound edge protection6 and gentamicin sponges4 to improve SSI rates following colorectal surgery mandate the investigation of novel techniques.

Initiated in the orthopaedic literature, a new technique of wound dressing has been described to reduce SSI. Incisional negative pressure wound therapy (NPWT) using devices such as the Prevena™ involves applying a wound vacuum sponge over a standard wound closure (including fascial closure and skin closure with staples). The incisional NPWT dressing is then left in place for 5 to 7 days before removal. A recent retrospective study by Bonds et al. described the ability of incisional NPWT to reduce SSI rates in open colorectal surgery from 29.3-12.5%.

The aim of the current study is to assess the clinical effectiveness of incisional NPWT to reduce SSI rates in open, re-operative colorectal surgery. The primary endpoint of this study is the occurrence of superficial SSI within 30 days after surgery and the secondary endpoints include, length of hospital stay and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* re-operative colorectal surgery
* excision or revision of prior anastomosis
* intestinal resection
* incisional hernia repair
* enterocutaneous fistula repair
* emergency settings

Exclusion Criteria:

* Laparoscopic or laparoscopic assisted procedures
* patients who had undergone a laparotomy within the preceding three months
* an active SSI at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2015-07; Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Liska, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sapci I, Camargo M, Duraes L, Jia X, Hull TL, Ashburn J, Valente MA, Holubar SD, Delaney CP, Gorgun E, Steele SR, Liska D. Effect of Incisional Negative Pressure Wound Therapy on Surgical Site Infections in High-Risk Reoperative Colorectal Surgery: A Randomized Controlled Trial. Dis Colon Rectum. 2023 Feb 1;66(2):306-313. doi: 10.1097/DCR.0000000000002415. Epub 2022 Apr 1. PMID 35358097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings
Started | 149 | 149
Completed | 149 | 149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings | Total
Number analyzed (Participants) | 149 | 149 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (16.4) | 52.2 (15.1) | 51 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 147
  Male | 75 | 76 | 151
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Superficial Surgical Site Infection
Description: Diagnosis will be based on criteria developed by the Centers for Disease Control (CDC)
Time Frame: within 30 days after the operation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings
Number analyzed (Participants) | 118 | 149
Participants
  Superficial Surgical Site Infection | 11 | 21
  No Superficial Surgical Site Infection | 107 | 128

2. Secondary Outcome: Length of Hospital Stay,
Description: number of days in hospital after surgery day
Time Frame: 30 days after operation
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings
Number analyzed (Participants) | 118 | 149
Days | 7 [5 to 9] | 6 [5 to 10]

3. Secondary Outcome: Cost Effectiveness
Description: ratio of costs between intervention and control group
Time Frame: 30 days after operation
Population: Study team ultimately decided not to collect this data
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Efficacy of the Device in Relation to the Degree of Contamination
Description: difference in SSI between groups
Time Frame: 30 days after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings
Number analyzed (Participants) | 149 | 149
Participants
  Clean-Contaminated | 15 | 12
  Contaminated | 94 | 90
  Dirty | 39 | 45
  No contamination | 1 | 2

ADVERSE EVENTS:
Time Frame: 30 days post surgery (+/- 7 days)
Arm/Group | Prevena™ Incisional NPWT | Standard Wound Dressings
All-Cause Mortality (participants affected / at risk) | 0/149 | 1/149
Serious Adverse Events (participants affected / at risk) | 11/149 | 19/149
Other Adverse Events (participants affected / at risk) | 92/149 | 84/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena™ Incisional NPWT (N=149) | Standard Wound Dressings (N=149)
Abcess (Infections and infestations) | 0 (0) | 1 (1)
Bladder Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Portal Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Altered mental status (Psychiatric disorders) | 0 (0) | 2 (2)
Reoperation (Surgical and medical procedures) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal Pain (General disorders) | 0 (0) | 2 (2)
Hyperglycemia (Investigations) | 0 (0) | 1 (1)
Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2)
Elevated Heart Rate (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 2 (2) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Internal Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ileostomy Ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena™ Incisional NPWT (N=149) | Standard Wound Dressings (N=149)
Ileus (Gastrointestinal disorders) | 22 (22) | 23 (23)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 12 (12)
Ureteric Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 9 (9)
Dehydration (General disorders) | 4 (4) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal Distension (General disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal Abscess (Infections and infestations) | 4 (4) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 5 (5)
Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Central Line bloodstream infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
High Ileostomy Output (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal Pain (General disorders) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Decreased Stoma output (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Drainage (General disorders) | 0 (0) | 2 (2)
Seroma/ Fluid Collection (General disorders) | 3 (3) | 3 (3)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2)
Malnutrition (Gastrointestinal disorders) | 1 (2) | 0 (0)
Reoperation due to stoma kinking (Surgical and medical procedures) | 1 (1) | 0 (0)
Elevated White Blood Cells (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Short Gut Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
C. Diff (Infections and infestations) | 1 (1) | 1 (1)
Mucosal Separation (General disorders) | 1 (1) | 1 (1)
Blood Clots from Stoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lightheadness (General disorders) | 1 (1) | 0 (0)
Enteritis (Infections and infestations) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Gas (General disorders) | 1 (1) | 0 (0)
Placement/ replacement of Lines/ Tubes (Surgical and medical procedures) | 2 (2) | 0 (0) — Includes PICC, NG tubes and PEG tubes
Leg Swelling (General disorders) | 1 (1) | 0 (0)
Increased Creatinine (Investigations) | 1 (1) | 0 (0)
Pancreatitis (Infections and infestations) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Wound Leak (General disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT02509260/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT02509260/ICF_001.pdf